CLINICAL TRIAL: NCT05119400
Title: Psychiatric Outcomes Following Inpatient Hospitalization For COVID-19
Brief Title: COVID-19 (Coronavirus Disease-2019) Psychiatric Outcomes
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit staff or funding to complete the study
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 20-08022609
Record Dates: First submitted 2021-10-27; First posted 2021-11-15 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Covid19; Anxiety; Mood; Cognitive Impairment
Keywords: Psychiatric Outcome; Inpatient Hospitalization
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 group: COVID-19 group will be made up of 30 patients that have a past diagnosis of COVID-19 with confirmed positive SARS-CoV-2 (Severe acute respiratory syndrome coronavirus 2) PCR (polymerase chain reaction) test in their electronic medical record and were previously hospitalized at NYP/WCM (NewYork Presbyterian/ Weill Cornell Medicine) between March 1 and December 31, 2020 for a minimum of three days.
  Administration of study instruments, including self-report measures of mood, anxiety, post-traumatic stress and adjustment, and objective neuropsychological tests of cognitive function will be done via telephone interview, videoconference interview, and/or Redcap survey for both groups.
- Comparison group: The subjects in comparison group will be 30 patients previously hospitalized at NYP/WCM between March 1 and December 31, 2020 for a minimum of three days. The recruited subjects would have undergone hospitalization secondary to a medical diagnosis that was not COVID-19.
  Administration of study instruments, including self-report measures of mood, anxiety, post-traumatic stress and adjustment, and objective neuropsychological tests of cognitive function will be done via telephone interview, videoconference interview, and/or Redcap survey for both groups.

SUMMARY:
The goal of this longitudinal and observational study is to better understand the psychiatric consequences of COVID-19 over time. Psychiatric outcomes like mood, anxiety, stress, and cognitive symptoms in patients who underwent inpatient hospitalization at NewYork-Presbyterian Hospital/Weill Cornell Medicine for COVID-19 will be assessed at 6 months or later post-discharge.

ELIGIBILITY:
Inclusion Criteria-COVID-19 group:

* Men and women age 18-89.
* Past diagnosis of COVID-19 with confirmed positive SARS-CoV-2 PCR test in electronic medical record
* English speaking
* Previously hospitalized at NYP/WCM between March 1 2020 and six months prior to enrollment for a minimum of three days.

Inclusion Criteria-Comparison group:

* Men and women age 18-89
* English speaking
* Previously hospitalized at NYP/WCM between March 1 2020 and six months prior to enrollment for a minimum of three days.
* Underwent hospitalization secondary to a medical diagnosis that was not COVID-19

Exclusion Criteria--COVID-19 group:

N/A

Exclusion Criteria--Comparison group:

* Past diagnosis of COVID-19
* Admitted to inpatient hospitalization due to, or past history of, a primary central nervous system relation etiology such as stroke, brain tumor, encephalitis, traumatic brain injury, multiple sclerosis, or Parkinson's disease.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients who were previously hospitalized at NYP/WCM between March 1 and December 31, 2020 for a minimum of three days will be enrolled.
  Out of 60, 30 patients would have a past diagnosis of COVID-19 and 30 patients would have undergone hospitalization secondary to a medical diagnosis that was not COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning as measured by Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) (English) | Once, 6 months to 36 months post-discharge from the hospital.
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) comprises auditory and visual subtasks of attention, language, visuospatial/constructional abilities, and immediate and delayed memory. Each subtask is assessed as accuracy (number of correct responses) and subsequently combined into a composite score (RBANS Total Scale score).

SECONDARY OUTCOMES:
Executive functioning as measured by the Oral Trail Making Test-B (OTMT-B; English) | Once, 6 months to 36 months post-discharge from the hospital.
  The oral version of the Trail Making Test (OTMT) assesses processing speed, working memory, and attention. Participants have to say out loud numbers and letters in alternating sequence and the time to completion is recorded.
Cognitive control as measured by the Stroop test (English) | Once, 6 months to 36 months post-discharge from the hospital.
  The Stroop Color and Word Test (SCWT) is used to assess verbal processing speed and ability to inhibit cognitive interference. Participants have to read out loud words, colors, and color words printed in different colored ink. The number of correct responses in 45 seconds is recorded.
Verbal intellectual ability as measured by the National Adult Reading Test (NART) for English speakers and the Word Accentuation Test (WAT). | Once, 6 months to 36 months post-discharge from the hospital.
  Participants have to read a set of words out loud and the number correct is recorded. Number of errors are recorded out of 61 words.
Verbal Fluency (English) | Once, 6 months to 36 months post-discharge from the hospital.
  This test requires participants to verbally produce words that start with given letters in a given time. The number of total valid words is used to indicate of successful selective information retrieval from memory.
Mood symptoms as assessed by DASS (English) | Once, 6 months to 36 months post-discharge from the hospital.
  Participants' moods will be assessed by Depression and Anxiety Scale (DASS) which is 42 item quantitative measure of three related negative emotional states of depression, anxiety and stress. The scores are interpreted for all three areas and higher scores indicate that the participant experiences increased emotional distress in either or all areas. For depression, the score ranges of 0-9 mean normal, 10-13 is mild, 14-20 moderate, 21-27 severe, and 28+ would be categorized under extremely severe depression. For anxiety, 0-7 is normal, 8-9 mild, 10-14 moderate, 15-19 severe, 20+ extremely severe. And for Stress, 0-14 is normal, 15-18 mild, 19-25 moderate, 26-33 severe, and 34+ extremely severe.
Mood symptoms as assessed by PANAS (English) | Once, 6 months to 36 months post-discharge from the hospital.
  The Positive and Negative Affect Schedule (PANAS) is a 20-item scale to measure affect. The scale consists of different words that alternate between positive and negative affect and each item is rated on a 5 point scale. Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Acceptance as assessed by AAQ-II (English) | Once, 6 months to 36 months post-discharge from the hospital.
  The Acceptance and Action Questionnaire (AAQ) is a 7-item self-report questionnaire used to measure psychological inflexibility and experiential avoidance. Scores range from 7- 49 with higher scores indicating higher level of inflexibility/avoidance.
Resilience as assessed by Brief Resilience Scale (English) | Once, 6 months to 36 months post-discharge from the hospital.
  The Brief Resilience Scale (BRS) is 6-item questionnaire used to assess the participant's perceived ability to recover from stressful events. The possible score range on each item is from 1 (low resilience) to 5 (high resilience).
Cognitive difficulties in daily life as assessed by Neuro Quality of Life (NeuroQOL) (English) | Once, 6 months to 36 months post-discharge from the hospital.
  NeuroQOL is a self-report questionnaires used to determine cognitive difficulties in participants' tasks of daily living. Scores range from 8-40 where lower score indicate that the participant experiences cognitive difficulties in their daily tasks and higher scores indicate minimum or no cognitive difficulties.
Cognitive function as assessed by Attention Network Test (ANT) | Once, 6 months to 36 months post-discharge from the hospital.
  ANT is a validated and computer-based paradigm that is based on an underlying attention/executive function network model of attention. It assesses three components of attention: alerting attention, orienting attention, and executive attention.
Cognitive function as assessed by EEG. | Once, 6 months to 36 months post-discharge from the hospital.
  An event-related potential (ERP) is the stereotypical voltage change that occurs in brain structures following specific cognitive events. When recorded using EEG, they are a powerful noninvasive method to study neural correlates of mental processes. We will record EEG while subjects engage in passive auditory cognitive processing and extract specific ERP components that are known to be sensitive to subtle cognitive weaknesses (N100, P300, N400).

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Jaywant, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification, will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to abj2006@med.cornell.edu. To gain access, requestors will need to sign data access agreement.